CLINICAL TRIAL: NCT05058677
Title: Aerosolized Endotracheal Lidocaine to Avoid Intracranial Pressure Spikes in Patients With Severe Traumatic Brain Injury
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: The University of Texas Health Science Center, Houston (Other)
Responsible Party: Principal Investigator, Thao L Nguyen, Assistant Professor, The University of Texas Health Science Center, Houston
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: HSC-MS-21-0254
Record Dates: First submitted 2021-09-16; First posted 2021-09-28 (Actual); Last update posted 2026-01-14 (Actual); Status verified 2026-01

CONDITIONS: Traumatic Brain Injury
Keywords: lidocaine; brain injury; intracranial pressure
MeSH Terms: conditions — Brain Injuries, Traumatic; Brain Injuries | interventions — Lidocaine; Sodium Chloride

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (6):
- aerosolized lidocaine then Instilled lidocaine solution then instilled saline solution (Experimental): Treatment will be performed before the endotracheal suctioning
  Interventions: Drug: aerosolized 2% lidocaine (20mg/ml); Drug: instilled 0.9% sodium chloride (NS); Drug: instilled 2% lidocaine solution; Procedure: Endotracheal Suctioning (ETS)
- aerosolized lidocaine then instilled saline solution then Instilled lidocaine solution (Experimental): Treatment will be performed before the endotracheal suctioning
  Interventions: Drug: aerosolized 2% lidocaine (20mg/ml); Drug: instilled 0.9% sodium chloride (NS); Drug: instilled 2% lidocaine solution; Procedure: Endotracheal Suctioning (ETS)
- Instilled lidocaine solution then aerosolized lidocaine then instilled saline solution (Experimental): Treatment will be performed before the endotracheal suctioning
  Interventions: Drug: aerosolized 2% lidocaine (20mg/ml); Drug: instilled 0.9% sodium chloride (NS); Drug: instilled 2% lidocaine solution; Procedure: Endotracheal Suctioning (ETS)
- Instilled lidocaine solution then instilled saline solution then aerosolized lidocaine (Experimental): Treatment will be performed before the endotracheal suctioning
  Interventions: Drug: aerosolized 2% lidocaine (20mg/ml); Drug: instilled 0.9% sodium chloride (NS); Drug: instilled 2% lidocaine solution; Procedure: Endotracheal Suctioning (ETS)
- Instilled saline solution then aerosolized lidocaine then Instilled lidocaine solution (Experimental): Treatment will be performed before the endotracheal suctioning
  Interventions: Drug: aerosolized 2% lidocaine (20mg/ml); Drug: instilled 0.9% sodium chloride (NS); Drug: instilled 2% lidocaine solution; Procedure: Endotracheal Suctioning (ETS)
- Instilled saline solution then Instilled lidocaine solution then aerosolized lidocaine (Experimental): Treatment will be performed before the endotracheal suctioning
  Interventions: Drug: aerosolized 2% lidocaine (20mg/ml); Drug: instilled 0.9% sodium chloride (NS); Drug: instilled 2% lidocaine solution; Procedure: Endotracheal Suctioning (ETS)

INTERVENTIONS:
Drug: aerosolized 2% lidocaine (20mg/ml) — The aerosolized solution to be used is 2% lidocaine (20 mg/ml) at a dose of 1.5 mg/kg with a maximum volume of 3 ml or adjusted to a volume of 3 ml with addition of NS solution.The aerosolized solution will be administered with an Aerogen ultrasonic nebulizer, which is standard of care for administering aerosolized solutions in our pediatric intensive care unit (PICU).After each treatment a 3-minute interval will be allowed prior to ETS and there will be a 4-6 hour wash out period between each treatment.
Drug: instilled 0.9% sodium chloride (NS) — The instilled solution will be given with a standard 3-5 ml syringe.After each treatment a 3-minute interval will be allowed prior to ETS and there will be a 4-6 hour wash out period between each treatment.
Drug: instilled 2% lidocaine solution — The instilled 2 % lidocaine solution used will be 1.5 mg/kg, with a max volume of 3 ml or adjusted to a volume of 3 ml with addition of NS solution.The instilled solution will be given with a standard 3-5 ml syringe.After each treatment a 3-minute interval will be allowed prior to ETS and there will be a 4-6 hour wash out period between each treatment.
Procedure: Endotracheal Suctioning (ETS) — ETS will be performed in a single pass using a closed-system suctioning. Suction will be applied only on withdrawal of the catheter and fraction of inspired oxygen (FIO2) will remain at 100% for 60 seconds following suctioning and then returned to the preprocedural level (baseline).

SUMMARY:
The purpose of this study is to evaluate the effectiveness of nebulized lidocaine before Endotracheal suctioning (ETS) compared to instilled lidocaine and the effectiveness of aerosolized lidocaine versus instilled normal saline before ETS in attenuating the increase of intracranial pressure (ICP) in severe head injured children and to evaluate the feasibility of a trial involving instilled lidocaine and aerosolized lidocaine for the management of ETS and to evaluate the safety of nebulized lidocaine in traumatic brain injury (TBI) compared to instilled lidocaine and instilled sodium chloride (NS).

ELIGIBILITY:
Inclusion Criteria:

* Patients admitted to the PICU of Memorial Hermann Children's Hospital
* Severe TBI with a Glasgow Coma Scale score 4-8
* Intubated and mechanically ventilated with an ICP monitor in place.
* Continuous invasive monitoring of arterial pressure
* Hemodynamically Stable, defined by normal blood pressure for age before the ETS. We will not exclude patients with norepinephrine to maintain goal blood pressures to maintain Cerebral perfusion pressure(CPP).

Exclusion Criteria:

* Patients with sustained ICP > 25 for more than 30 minutes mm Hg despite medical or neurosurgical intervention
* Moderate/Severe Acute respiratory distress syndrome (ARDS) with an oxygenation index > 8
* Pulmonary hemorrhage
* Patients receiving neuromuscular blockade
* Use of other vasopressors for other causes of shock (cardiogenic, hypovolemic and septic)

Max Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 10 (Actual)
Dates: Start 2021-11-09 (Actual); Primary Completion 2025-06-30 (Actual); Study Completion 2025-06-30 (Actual)

PRIMARY OUTCOMES:
Maximum difference between baseline ICP and highest ICP levels as measured by the ICP monitor in instilled lidocaine versus nebulized lidocaine | from baseline to upto 15 minutes after ETS
  A Codman Intraparenchymal Catheter will measure the ICP.The ICP will be transduced and measured numerically and continuously in real time on the patient's bedside monitor.

SECONDARY OUTCOMES:
Maximum difference between baseline ICP and highest ICP levels as measured by the ICP monitor in nebulized lidocaine and normal saline | from baseline to up to 15 minutes after ETS
  A Codman Intraparenchymal Catheter will measure the ICP.The ICP will be transduced and measured numerically and continuously in real time on the patient's bedside monitor.
Number of patients with worsening respiratory dynamics | from baseline to up to 15 minutes after ETS
  This will be measured by increasing oxygenation index or worsening compliance, measured by any increase in the peak pressure for volume ventilated patients.

CONTACTS AND LOCATIONS:
Overall Officials: Thao L Nguyen, DO, FAAP, Principal Investigator — The University of Texas Health Science Center, Houston
Locations (1):
- The University of Texas Health Science Center at Houston, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: No